CLINICAL TRIAL: NCT04206956
Title: Anxiety and Chronic Postsurgical Pain Following Ambulatory Surgery in Children
Acronym: ANXIDOU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Saint-Brieuc (Other)
Responsible Party: Sponsor
Other Study IDs: CHSB-2019-05-P2-ANXIDOU
Record Dates: First submitted 2019-12-09; First posted 2019-12-20 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Ambulatory Surgery; Children, Only; Inguinal Hernia; Umbilical Hernia; Urologic Surgery
Keywords: pediatric department; children; chronic postsurgical pain; perioperative anxiety
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Umbilical; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, monocentric, observationnal study. The primary objective of this study is to identify if presurgical child or/and parental anxiety is predictive of chronic postsurgical pain in abdominal or urologic ambulatory surgery.

DETAILED DESCRIPTION:
The post surgical pain guidelines recommend to identify predictive factors, especially for vulnerable subjects.

For children, there is few data about predictive factors of postoperative pain after ambulatory surgery.

The objective of this study is to collect preoperative data (preoperative children's anxiety and parental anxiety) and postoperative data (postoperative pain measure: the day of surgery and 3 months after surgery) for children undergoing abdominal ou urologic ambulatory surgery, and to determine if there is a relationship between these data (Odds Ratio)

ELIGIBILITY:
Inclusion Criteria:

* child from 3 to 18 years old
* undergoing scheduled urology or abdominal ambulatory surgery
* child and parents speaking French
* affiliation to national health insurance

Exclusion Criteria:

* emergency surgery
* lack of parents consent
* no parental support on surgery day

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing scheduled abdominal or urologic ambulatory surgery
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Children's preoperative anxiety | Preoperative : day of surgery
  - For children younger than 12 : mYPAS (the Modified Yale Preoperative Anxiety Scale).
  If the score is less than 24 : quiet child. If the score is greater than 24 : anxious child
  - For children older than 12 : anxiety visual analog scale (VAS) From 0 (better) to 10 (worse)
Parents' preoperative anxiety | Preoperative: day of surgery
  anxiety visual analog scale (VAS) From 0 (better) to 10 (worse). More than 3/10 means "anxious"
children's pain | postoperative: day of surgery
  * for children younger than 6: Evendol scale. From 0 (better) to 15 (worse)
  * for children older than 6: anxiety visual analog scale (VAS) From 0 (better) to 10 (worse).
Chronic postsurgical pain in children | 3 months after surgery
  For all children, score PPMP (Postoperative Pain Measure for Parents) From 0 (better) to 10 (worse)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Barbarot, Dr, Principal Investigator — Centre Hopsitalier Saint-Brieuc
Locations (1):
- Centre Hospitalier de Saint-Brieuc, Saint-Brieuc, France

REFERENCES:
- [Background] Rabbitts JA, Fisher E, Rosenbloom BN, Palermo TM. Prevalence and Predictors of Chronic Postsurgical Pain in Children: A Systematic Review and Meta-Analysis. J Pain. 2017 Jun;18(6):605-614. doi: 10.1016/j.jpain.2017.03.007. Epub 2017 Mar 29. PMID 28363861
- [Background] Batoz H, Semjen F, Bordes-Demolis M, Benard A, Nouette-Gaulain K. Chronic postsurgical pain in children: prevalence and risk factors. A prospective observational study. Br J Anaesth. 2016 Oct;117(4):489-496. doi: 10.1093/bja/aew260. Epub 2016 Oct 17. PMID 28077537
- [Background] Noel M, Rosenbloom B, Pavlova M, Campbell F, Isaac L, Page MG, Stinson J, Katz J. Remembering the pain of surgery 1 year later: a longitudinal examination of anxiety in children's pain memory development. Pain. 2019 Aug;160(8):1729-1739. doi: 10.1097/j.pain.0000000000001582. PMID 31335643
- [Background] Chieng YJ, Chan WC, Klainin-Yobas P, He HG. Perioperative anxiety and postoperative pain in children and adolescents undergoing elective surgical procedures: a quantitative systematic review. J Adv Nurs. 2014 Feb;70(2):243-55. doi: 10.1111/jan.12205. Epub 2013 Jul 19. PMID 23865442
- [Background] Page MG, Campbell F, Isaac L, Stinson J, Katz J. Parental risk factors for the development of pediatric acute and chronic postsurgical pain: a longitudinal study. J Pain Res. 2013 Sep 30;6:727-41. doi: 10.2147/JPR.S51055. eCollection 2013. PMID 24109194
- [Background] Rabbitts JA, Zhou C, Groenewald CB, Durkin L, Palermo TM. Trajectories of postsurgical pain in children: risk factors and impact of late pain recovery on long-term health outcomes after major surgery. Pain. 2015 Nov;156(11):2383-2389. doi: 10.1097/j.pain.0000000000000281. PMID 26381701
- [Background] Birnie KA, Chorney J, El-Hawary R; PORSCHE Study Group. Child and parent pain catastrophizing and pain from presurgery to 6 weeks postsurgery: examination of cross-sectional and longitudinal actor-partner effects. Pain. 2017 Oct;158(10):1886-1892. doi: 10.1097/j.pain.0000000000000976. PMID 28598902
- [Background] Kristensen AD, Ahlburg P, Lauridsen MC, Jensen TS, Nikolajsen L. Chronic pain after inguinal hernia repair in children. Br J Anaesth. 2012 Oct;109(4):603-8. doi: 10.1093/bja/aes250. Epub 2012 Jul 24. PMID 22831892
- [Background] Mossetti V, Boretsky K, Astuto M, Locatelli BG, Zurakowski D, Lio R, Nicoletti R, Sonzogni V, Maffioletti M, Vicchio N, Ivani G. Persistent pain following common outpatient surgeries in children: A multicenter study in Italy. Paediatr Anaesth. 2018 Mar;28(3):231-236. doi: 10.1111/pan.13321. Epub 2018 Jan 20. PMID 29352738
- [Background] Pinto PR, McIntyre T, Nogueira-Silva C, Almeida A, Araujo-Soares V. Risk factors for persistent postsurgical pain in women undergoing hysterectomy due to benign causes: a prospective predictive study. J Pain. 2012 Nov;13(11):1045-57. doi: 10.1016/j.jpain.2012.07.014. Epub 2012 Oct 12. PMID 23063345